CLINICAL TRIAL: NCT06372756
Title: Evaluation of Deep Learning Reconstruction Algorithms in Dual Low-dose CT Vascular Imaging
Brief Title: Deep Learning Reconstruction Algorithms in Dual Low-dose CTA
Status: Recruiting | Type: Observational
Sponsor: Hao Tang (Other)
Responsible Party: Sponsor-Investigator, Hao Tang, associate chief physician, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 102122
Record Dates: First submitted 2024-04-11; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Deep Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard dose group: Raw data from 400 patients with conventional dose head and neck CTA, coronary CTA, and abdominal CTA were included. Filtered back-projection, iteration, and deep learning reconstruction were performed. To evaluate the impact of deep learning reconstruction on image quality and diagnostic performance in patients with conventional dose CTA.
  Interventions: Diagnostic Test: Deep learning image reconstruction
- Double low dose group: Raw data from 800 patients with low tube voltage and contrast medium head and neck CTA, coronary CTA, and abdominal CTA were included. Filtered back-projection, iteration, and deep learning reconstruction were performed. To evaluate the impact of deep learning reconstruction on image quality and diagnostic performance in patients with double-low-dose CTA.
  Interventions: Diagnostic Test: Deep learning image reconstruction

INTERVENTIONS:
Diagnostic Test: Deep learning image reconstruction — Deep learning image reconstruction (DLIR) is a newly developed artificial intelligence noise reduction algorithm in recent years. It trains massive high-quality FBP data sets to learn to distinguish noise and signal, so as to selectively reduce noise and reconstruct high-quality images with low-quality image data.

SUMMARY:
The goal of this observational study is to evaluate the impact of deep learning image reconstruction on the image quality and diagnostic performance of double low-dose CTA. The main question it aims to answer is to explore the feasibility of deep learning image reconstruction in double low-dose CTA.

DETAILED DESCRIPTION:
1. The raw data from patients who underwent head and neck CTA, coronary CTA, and abdominal CTA in both standard dose and double low-dose groups were included.
2. Techniques such as filtered back projection, iterative reconstruction, and deep learning reconstruction were performed.
3. The feasibility of deep learning reconstruction in double low-dose CTA was evaluated based on image quality and diagnostic performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck CTA, coronary artery CTA, and abdominal CTA due to stroke, coronary heart disease and abdominal inflammatory disease, and abdominal tumors.

Exclusion Criteria:

* Age <18 years, pregnancy, allergic reaction to iodine contrast agent, renal insufficiency, and severe hyperthyroidism.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy or diseased adults undergoing CT vascular imaging
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The specificity and sensitivity calculated through the optimal cutoff value of the receiver operating characteristic curve. | 2026.1
  The specificity and sensitivity were calculated separately for the standard dose group and the double low-dose group using the optimal cutoff value from the receiver operating characteristic curve, for the purpose of comparing diagnostic accuracy between the two groups.

SECONDARY OUTCOMES:
The signal-to-noise ratio calculated from image CT values and noise | 2026.1
  The signal-to-noise ratio was calculated separately for the standard dose group and the double low-dose group using image CT values and noise, to assess the image quality between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Tang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
To protect the participant privacy, the relevant data is not shared until the participants' consent